CLINICAL TRIAL: NCT02653833
Title: Skeletal Muscle Blood Flow in Becker Muscular Dystrophy
Brief Title: The Study of Skeletal Muscle Blood Flow in Becker Muscular Dystrophy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI passed away
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00041688
Record Dates: First submitted 2015-12-14; First posted 2016-01-12 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-06

CONDITIONS: Muscular Dystrophy
Keywords: Becker; Muscular Dystrophy; Skeletal Muscle; blood flow; Ultrasound
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Controls (HC) (Experimental): Healthy men currently taking no medications will be asked to perform graded hand-grip exercise while a contrast enhanced ultrasound (CEU) probe is placed over their forearm to measure blood flow. This is repeated at baseline and shortly after taking beetroot juice extract.
  Interventions: Drug: Tadalafil 20 MG; Other: beetroot juice extract
- Becker Muscular Dystrophy (BMD) (Experimental): currently taking no medications will be asked to perform graded hand-grip exercise while a contrast enhanced ultrasound (CEU) probe is placed over their forearm to measure blood flow. Using a lower body negative pressure (LBNP) chamber, the subjects are tested for impaired exercise induced vasodilation to the skeletal muscle or "functional sympatholysis". This is repeated at baseline and shortly after taking beetroot juice extract.
  Interventions: Drug: Tadalafil 20 MG; Other: beetroot juice extract

INTERVENTIONS:
Drug: Tadalafil 20 MG — Blood flow to the forearm is visualized via an ultrasound technique at rest and with graded exercise. The experiment is then repeated shortly after the subject takes the study agent, beetroot juice extract.
Other: beetroot juice extract — Blood flow to the forearm is visualized via an ultrasound technique at rest and with graded exercise. The experiment is then repeated shortly after the subject takes the study agent, beetroot juice extract.

SUMMARY:
This pilot study tests the hypothesis that the medication nitric oxide extract from beetroot juice improves blood flow to the skeletal muscle during exercise. The investigators will use cutting edge technology with contrast enhanced ultrasound to visualize the microvascular blood supply to the forearm. Animal studies have shown reversal of muscle damage with improved delivery of blood to the exercising muscle. This research aims to understand the mechanism of action of this medication in a way it has never been studied before. The results may help benefit individuals with muscular Dystrophy in the future.

DETAILED DESCRIPTION:
The subjects are asked to perform a graded hand-grip exercise while blood flow to the skeletal muscle is visualized by contrast enhanced ultrasound.

This is done at baseline and after taking the study agent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man, aged 18 to 45 years, currently taking no medication. OR
* Clinical diagnosis of Becker Muscular Dystrophy (BMD), aged 18 to 45 years, and currently taking no medication.

Exclusion Criteria:

* Hypertension, diabetes, heart failure, liver disease
* ECG evidence of prolonged QT interval

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Blood Flow | At baseline and within one hours after taking beetroot juice or Tadalafil
  Exercise induced skeletal muscle perfusion is measured by contrast-enhanced ultrasound (CEU) during graded voluntary contraction on a hand grip dynamometer.

SECONDARY OUTCOMES:
Change in Measured Functional Sympatholysis | At baseline, and within an hour after taking beetroot juice or Tadalafil
  Functional sympatholysis (attenuation of exercise induced skeletal muscle vasoconstriction) is assessed using a lower body negative pressure chamber.
Change in Measured Flow Mediated Dilation (FMD) | At baseline, and within an hour after taking beetroot juice or Tadalafil
  Endothelial function is assessed by measuring flow-mediated dilation (FMD) by Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No